CLINICAL TRIAL: NCT03719339
Title: Validating Injury to Renal Transplant Using Urinary Signatures in Children
Brief Title: VIRTUUS Children's Study
Acronym: VIRTUUS
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-013841; 1R01HD091185-01 (NIH)
Record Dates: First submitted 2018-07-13; First posted 2018-10-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Renal Transplant Rejection; Pediatric Kidney Disease; End Stage Renal Disease; Nephropathy; BK Virus (Nephropathy); Antibody-mediated Rejection; Acute Cellular Graft Rejection
Keywords: Kidney disease; Kidney allograft
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, sputum, urine, tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

SUMMARY:
The objective of the VIRTUUS Children's Study is to adapt identified and validated adult noninvasive diagnostic and prognostic biomarkers for the characterization of allograft status in pediatric recipients of kidney allografts.

DETAILED DESCRIPTION:
Advances in immunosuppressive regimens have significantly improved short-term allograft survival for kidney transplant recipients. Yet, long-term allograft survival remains static. For children with end-stage renal disease (ESRD), improvements in long-term outcomes are greatly needed. Children with ESRD require multiple transplants over a lifetime, incurring repeated surgical and immunological risks with each newly transplanted organ. Allograft injury occurs primarily due to acute cellular rejection (ACR) and/or antibody mediated rejection (AMR) and viral infections, such as BK virus associated nephropathy (BKVN). A major hindrance to promoting long-term allograft survival is the lack of non-invasive diagnostic and prognostic biomarkers to reliably detect early injury in the allograft before clinical manifestations arise.

The incidence of acute rejection (AR) in children in the first year post-transplant is 10-13%[1]. The current gold standard for diagnosing AR is core needle biopsy; however, biopsy is highly invasive, incurs risk of bleeding and graft loss, is subject to sampling error and lacks sensitivity and specificity for early injury. Since immune responses are dynamic over time, single biopsies do not adequately capture anti-allograft immunity, but repeat biopsies are impractical in children who often require sedation and hospitalization for biopsies. Other markers, such as serum creatinine, have low sensitivity and specificity for early kidney allograft damage.

The ability to identify sub-clinical kidney allograft injury using minimally invasive, robust, biomarkers with high sensitivity and specificity in pediatric recipients would represent a major advance in pediatric kidney transplant care. In the Clinical Trials in Organ Transplantation (CTOT)-04 study, a NIH-sponsored, multicenter, prospective study of adult kidney allograft recipients, members of the VIRTUUS team were able to diagnose and predict ACR using urinary cell mRNA and metabolite profiles with high sensitivity and specificity[2, 3]. In addition, the investigators validated a urinary cell mRNA signature that distinguishes acute rejection (AR) from acute tubular injury (ATI) and ACR from AMR as well as a urinary cell mRNA signature diagnostic and prognostic of BKVN[3-5]. The overarching objective of this VIRTUUS proposal is to adapt existing validated adult noninvasive diagnostic and prognostic biomarkers to characterize allograft status in pediatric recipients of kidney allografts. Specifically, the investigators will investigate 1) whether the adult urinary cell 3-gene signature is diagnostic and prognostic of ACR in pediatric recipients of kidney allografts, 2) whether the combined metabolite and the urinary cell 3-gene signature is diagnostic and prognostic of ACR in pediatric recipients of kidney allografts, 3) whether levels of BKV VP-1 mRNA in urinary cells are diagnostic of BKVN, and 4) whether urinary cell levels of plasminogen activator inhibitor -1 (PAI-1) mRNA and serum creatinine levels predict allograft failure.

Investigators propose to validate early immunologic markers that have shown to be prognostic and diagnostic in adult kidney transplant recipients in pediatric kidney transplant recipients. Investigator findings will significantly advance the field of pediatric transplantation by moving toward proactive, tailored immunosuppressive regimens that minimize morbidity and optimize long-term allograft survival.

The Investigator's primary objective is to hypothesize that: (i) the adult urinary cell 3-gene signature will be diagnostic and prognostic of ACR in longitudinally collected urine samples from children with kidney transplants; and (ii) combined metabolite and mRNA biomarkers have greater ability to diagnose ACR than the mRNA or metabolite signature alone and (iii) levels of BKV VP-1 mRNA are diagnostic of BK virus nephropathy (BKVN) and (iv) urinary cell levels of plasminogen activator inhibitor-1 (PAI-1) mRNA and serum creatinine levels predict allograft failure.

Investigators seek to:

1. Determine if the adult urinary cell 3-gene signature is diagnostic and prognostic of ACR in pediatric kidney allograft recipients,
2. Evaluate whether a combined metabolite and the 3-gene urinary mRNA signature is diagnostic and prognostic of ACR and
3. Test the hypothesis that BKV-VP-1 mRNA levels in urinary cells are diagnostic of BKVN, and to test the hypothesis that a two variable prediction model composed of urinary cell level of PAI-1 mRNA and serum creatinine levels, both measured at the time of BKVN biopsy diagnosis, predict future graft failure

Secondary objectives include the following:

1. Create a repository of DNA samples from urine, saliva, discarded blood and tissue, and deceased donor blood and tissue to use for future research studies that will examine genome-wide associations with rejection and viral infections in pediatric kidney transplant recipients and
2. Create a biobank of samples of left-over blood and deceased donor blood to later examine associations between urine and blood proteomics and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 2 to 18 years at the time of recruitment
* Receiving the first, or additional, incident kidney transplants.
* Have an existing/prevalent transplant with a scheduled kidney allograft biopsy.
* Parental/guardian permission (informed consent) and, if appropriate, child assent.

Exclusion Criteria:

• Patient's primary medical team feels the subject's participation is not safe.

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Subjects 2 to 18 years of age meeting inclusion criteria will be recruited from the participating sites' Nephrology outpatient clinics or inpatient settings. All sites may choose to enroll Spanish speaking subjects pending the site has necessary resources to translate/interpret study related information. Sites choosing to enroll Spanish speaking subjects will have a native speaking translator or interpreter available to prevent any miscommunication during the consent process.
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Amount of CD3E mRNA (CD3-epsilon polypeptide) | 48 months
  The amount of mRNA observed in urinary sample biopsy.
Amount of CXCL10 (chemokine C-X-C motif ligand 10) | 48 months
  The amount of mRNA observed in urinary sample biopsy.
Amount of 18s rRNA | 48 months
  The amount of mRNA observed in urinary sample biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Keating, DPhil, Principal Investigator — Children's Hospital of Philadelphia and Hospital of The University of Pennsylvania
Locations (13):
- United States (12):
  - University of California-San Diego, Rady Children's Hospital, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Joan & Sanford I. Weill Medical College of Cornelle University, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - CHOP, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Vancouver Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Ettenger RB, Seifert ME, Blydt-Hansen T, Briscoe DM, Holman J, Weng PL, Srivastava R, Fleming J, Malekzadeh M, Pearl M. Detection of Subclinical Rejection in Pediatric Kidney Transplantation: Current and Future Practices. Pediatr Transplant. 2024 Sep;28(6):e14836. doi: 10.1111/petr.14836. PMID 39147695